CLINICAL TRIAL: NCT06975748
Title: A Phase II, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety and Efficacy of STSP-0902 Ophthalmic Solution in Patients With Neurotrophic Keratitis
Brief Title: A Phase II Study of STSP-0902 Ophthalmic Solution in Patients With Neurotrophic Keratitis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSP-0902-02-002
Record Dates: First submitted 2025-04-15; First posted 2025-05-16 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Neurotrophic Keratitis
Keywords: STSP-0902; Ophthalmic Solution; Neurotrophic Keratitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose 3 Times Daily Arm (Experimental): Low dose of STSP-0902 ophthalmic solution to the affected eye(s), 3 times daily for 8 weeks
  Interventions: Drug: STSP-0902 ophthalmic solution
- Low Dose 6 Times Daily Arm (Experimental): Low dose of STSP-0902 ophthalmic solution to the affected eye(s), 6 times daily for 8 weeks
  Interventions: Drug: STSP-0902 ophthalmic solution
- High Dose 3 Times Daily Arm (Experimental): High dose of STSP-0902 ophthalmic solution to the affected eye(s), 3 times daily for 8 weeks
  Interventions: Drug: STSP-0902 ophthalmic solution
- Control Arm (Placebo Comparator): STSP-0902 Placebo to the affected eye(s), 3 or 6 times daily for 8 weeks
  Interventions: Drug: STSP-0902 Placebo

INTERVENTIONS:
Drug: STSP-0902 ophthalmic solution — Eye drop, 3 times daily for 8 weeks
  Arms: High Dose 3 Times Daily Arm; Low Dose 3 Times Daily Arm
Drug: STSP-0902 ophthalmic solution — Eye drop, 6 times daily for 8 weeks
  Arms: Low Dose 6 Times Daily Arm
Drug: STSP-0902 Placebo — Eye drop, 3 or 6 times daily for 8 weeks
  Arms: Control Arm

SUMMARY:
This is a Phase II, double-blind, placebo-controlled study to evaluate the safety and efficacy of STSP-0902 ophthalmic solution in patients with neurotrophic keratitis (NK). The study plans to enroll 48 patients with Mackie Stage 2 or 3 NK affecting one or both eyes. Eligible subjects will be randomized 1:1:1 into three dosing groups. Each dosing group will follow a drug-placebo allocation (12 active: 4 placebo). Treatment involves topical ocular administration for 8 weeks. Subjects who are not healed after the 8 weeks of masked treatment period will be permitted to receive standard of care during the follow-up period

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged between 18 to 80 years (inclusive).
2. Diagnosed with NK in one or both eyes, with the study eye classified as Mackie Stage 2 (PED) or Stage 3 (corneal ulcer), and with a maximum corneal defect diameter ≥2 mm.
3. Reduced or absent corneal sensitivity in the defect area and at least 1 adjacent corneal quadrant, confirmed by: ≤40 mm using the aesthesiometer or cotton swab test demonstrating marked reduction or absence of corneal sensitivity.
4. NK duration >2 weeks in the study eye, as confirmed by the investigator based on medical history.
5. No improvement in the study eye for ≥7 days prior to randomization.
6. Effective non-pharmacological contraception used by the subject (and partner, if applicable) throughout the trial and for 3 months after the last dose, with no plans for pregnancy or gamete donation.
7. Voluntarily sign informed consent, with willingness and ability to comply with study procedures, follow-ups, and assessments.

Exclusion Criteria:

1. Any eye with corneal stromal ulceration involving >1/3 of corneal thickness or at risk of corneal melting/perforation.
2. Active infection (bacterial, viral, fungal, amoebic, chlamydial) in any eye, or active ocular inflammation unrelated to NK.
3. Study eye with other ocular diseases requiring topical medication during the trial.
4. Bilateral vision loss severely impacting daily life, as assessed by the investigator.
5. Study eye with Schirmer I test ≤3 mm/5 minutes.
6. Severe lagophthalmos, eyelid margin disease, or meibomian gland dysfunction in the study eye that may impair corneal healing or trial outcomes.
7. Study eye with any surgery within 3 months prior to randomization (including corneal/non-corneal surgeries affecting trial assessments, except surgeries related to NK etiology), or planned ocular surgery during the trial.
8. Study eye with prior surgical intervention for NK (e.g., tarsorrhaphy, conjunctival flap) that may confound efficacy assessments, or amniotic membrane transplantation within 6 weeks prior to randomization.
9. Study eye with botulinum toxin injections to the levator muscle within 3 months prior to randomization or planned during the trial.
10. Requirement to wear contact lenses during the trial.
11. History of inefficacy or poor response to nerve growth factor (NGF) eye drops in any eye.
12. Use of autologous serum eye drops, deproteinized calf blood extracts, or other growth factor-containing ocular medications in the study eye within 3 days prior to randomization or planned during the trial.
13. Use of NSAIDs, corticosteroids, or immunosuppressive eye drops in the study eye within 1 week prior to randomization or planned during the trial.
14. Use of neurotoxic drugs (e.g., antipsychotics, antiepileptics, antihistamines) or systemic immunosuppressants within 4 weeks prior to randomization or planned during the trial.
15. Poorly controlled systemic or ocular conditions (e.g., diabetic retinopathy, uveitis, autoimmune diseases, malignancies, psychiatric disorders) that may confound efficacy assessments or compliance, as judged by the investigator.
16. Known hypersensitivity to the study drug, its excipients, or components of trial-related ophthalmic tests (e.g., fluorescein).
17. History of drug abuse or alcohol dependence.
18. Participation in another interventional trial (drugs, devices, or vaccines) within 3 months prior to randomization or planned during this trial.
19. Female subjects who are pregnant, breastfeeding, or test positive for serum pregnancy; or who are failure to use effective contraception for 2 weeks prior to screening, during the trial, or for 3 months post-dosing.
20. Difficulty administering eye drops, venous blood sampling, or history of needle phobia/vasovagal syncope.
21. Any other condition deemed unsuitable for trial participation by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Screening to Week 10
  Number of participants with ocular and systemic adverse events as assessed by CTCAE v5.0.
Ocular Symptoms and Signs | Screening to Week 10
  Number of subjects with clinically significant changes in ocular symptoms and signs.
Intraocular Pressure (IOP) Measurements | Screening to Week 10
  Change in IOP is measured using a non-contact tonometer (In cases requiring precise IOP evaluation, a contact tonometer may be used).
Slit-Lamp Examinations | Screening to Week 10
  Number of subjects with clinically significant changes detected by slit-lamp microscope. The slit lamp examinations will encompass the eyelids, conjunctiva, cornea, anterior chamber, aqueous humor, iris, lens, and other relevant ocular structures.
Optical Coherence Tomography (OCT) Results | Screening to Week 10
  Proportion of corneal thickness affected by the stromal ulceration, as evaluated by the investigator.
Clinically Significant Changes in Vital Signs | Screening to Week 10
  Vital signs include body temperature in ℃, pulse rate in bpm, respiration rate in breaths/ minute, and blood pressure in mmHg.
Clinically Significant Changes in Physical Examinations | Screening to Week 10
  Physical examinations include assessments of general status, skin and mucous membranes, lymph nodes, head and neck, chest, abdomen, musculoskeletal system, spine/extremities, nervous system, and additional regions as clinically indicated.
Clinically Significant Changes in 12-Lead ECGs | Screening to Week 10
  Parameters measured: Heart rate in bpm, P-R interval in ms, QRS duration in ms, QT interval in ms, QTc interval in ms.
Clinically Significant Laboratory Abnormalities | Screening to Week 10
  Blood samples will be collected for hematology, blood biochemistry and coagulation function. Urine sample will be collected for and urinalysis.

SECONDARY OUTCOMES:
Corneal Healing | Baseline to Week 10
  Percentage of subjects achieving corneal healing assessed via corneal fluorescein staining by the investigator
Corneal Sensitivity | Baseline to Week 10
  Evaluation of sensation in corneal quadrants using the aesthesiometer
Patients with Deterioration | Baseline to Week 10
  Percentage of Subjects with Disease Deterioration
Best Corrected Visual Acuity (BCVA) | Baseline to Week 8
  Change in BCVA from Baseline
Tear Secretion | Baseline to Week 8
  Change in Tear Secretion from Baseline as evaluated via Schirmer I test
Visual Quality of Life Assessed Using the NEI-VFQ-25 | Baseline to Week 8
  VFQ-25 is a questionnaire composed of 25 vision-targeted questions assessing 11 vision-related constructs, along with a single-item question to rate general health. Original responses from the questionnaire are recoded to a scale ranging from 0 to 100, where a higher score indicates better visual function. Each question corresponds to one of the 12 sub-scales and scores for each sub-scale are calculated by averaging its constituent questions. The overall composite score is generated by averaging the 11 vision-specific sub-scales, excluding the general health item.
STSP-0902 concentration | Baseline to Week 10
  Measurement of STSP-0902 in plasma after drug administration
Incidence of positive detection of anti-STSP-0902 antibodies | Baseline to Week 10
  Measurement of anti-drug antibody (ADA) to STSP-0902 in plasma after drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Shi, Ph.D, Principal Investigator — Shandong First Medical University Affiliated Eye Hospital; Ting Wang, Ph.D, Principal Investigator — Shandong First Medical University Affiliated Eye Hospital
Locations (1):
- Shandong First Medical University Affiliated Eye Hospital, Jinan, Shandong, China